CLINICAL TRIAL: NCT06738147
Title: "Effect of Pelvic Floor Muscle Training on Postural Balance and Fall Risk in Postmenopausal Females With Urinary Incontinence"
Brief Title: Effect of Pelvic Floor Muscle Training on Balance and Fall Risk in Females With Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hager Mohey Eldien Abdel Aziz Mahmoud, Assistant lecturer of physical therapy for woman health at deraya university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P.T.REC/012/005377
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence; Balance
Keywords: pelvic floor; postural balance; fall risk; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (A) (Experimental): It will consist of (15) postmenopausal females are complaining of urinary incontinence and balance disturbances who will be treated by pelvic floor muscle training (PFMT) for 30 min., 3 sessions/ week in addition to traditional physical and balance training program (proprioception training and balance exercises for the static and dynamic components of balance for 30 min., three sessions/ week for six weeks.
  Interventions: Other: pelvic floor muscle training; Other: balance exercises
- Control Group (B) (Other): It will consist of (15) postmenopausal females are complaining of urinary incontinence and balance disturbances who will be treated by traditional physical and balance training program only (proprioception training and balance exercises for the static and dynamic components of balance for 30 min., three sessions/ week for six weeks.
  Interventions: Other: balance exercises

INTERVENTIONS:
Other: pelvic floor muscle training — pelvic floor muscle training (PFMT) for 30 min., 3 sessions/ week in addition to traditional physical and balance training program (proprioception training and balance exercises for the static and dynamic components of balance for 30 min., three sessions/ week for six weeks.
  Other Names: balance exercises
  Arms: Experimental Group (A)
Other: balance exercises — traditional physical and balance training program (proprioception training and balance exercises for the static and dynamic components of balance for 30 min., three sessions/ week for six weeks.

SUMMARY:
Understanding the relationship between Pelvic floor muscle dysfunctions as stress urinary incontinence with Postural balance ability and subsequent fall risk in postmenopausal females is important in terms of injury prevention and decrease morbidity and mortality rate among postmenopausal females. Therefore, this study investigating the effect of pelvic floor muscle training on postural balance and fall risk in postmenopausal females with stress urinary incontinence.

DETAILED DESCRIPTION:
Thirty post-menopausal females will participate in this study. They will be selected from the outpatient clinic at Daraya University.They will be randomly assigned in two groups experimental (A) and control (B) group, each group will have (15) postmenopausal female. Experimental Group (A):

It will consist of (15) postmenopausal females are complaining of urinary incontinence and balance disturbances who will be treated by pelvic floor muscle training (PFMT) for 30 min., 3 sessions/ week in addition to traditional physical and balance training program (proprioception training and balance exercises for the static and dynamic components of balance for 30 min., three sessions/ week for six weeks.

Control Group (B):

It will consist of (15) postmenopausal females are complaining of urinary incontinence and balance disturbances who will be treated by traditional physical and balance training program only (proprioception training and balance exercises for the static and dynamic components of balance for 30 min., three sessions/ week for six weeks.

All females in both groups will be evaluated for urinary incontinence through ultrasonography and pelvic floor bother questionnaire (PFBQ) at the beginning of the study and at the end of treatment period. Also, static, and dynamic balance performance and fall risk will be assessed in the beginning of the study and at the end of treatment period through the Biodex balance system and Tinetti Performance Oriented Mobility Assessment (POMA). All participants will be given an explanation of study protocol, and an informed consent form will be signed by each female

ELIGIBILITY:
Inclusion Criteria:

* 1. All females will be postmenopausal. 2. Their ages will range from: 50-60 years. 3. Their BMI will be less than 30 kg\m2. 4. All females will be suffering from urinary incontinence. 5. All females will be sedentary. 6. All females will have balance disorders. 7.All females will be able to walk across a small room without an assistive device.

Exclusion Criteria:

1. History of lower extremity injury, surgery or pain during ADL.
2. Females having any vestibular problems, otitis media, labyrinthitis or any inner ear problems that affect balance.
3. Women with mild, moderate and severe cognitive deficits.
4. Women with neurological diseases, including conditions after a Stroke.
5. Females with a history of brain injury.
6. Females with significant visual and hearing damage confirmed by neurological examination.
7. Females with serious internal orthopedic and oncological diseases.

   -

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
pelvic floor muscle activity | 3 months
  Assessment of pelvic floor muscle by Ultrasound imaging device, it will be used to assess PFM activity by measuring bladder base displacement (as a marker for PFM activity)
antero posterior stability index | 3 months
  Indicator for dynamic postural stability
Medio lateral stability index | 3 months
  Indicator for dynamic postural stability
Overall stability index | 3 months
  Indicator for dynamic postural stability
stability an sway indexes | 3 months
  Indicator for fall risk

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF